# Foundation Fighting Blindness (FFB) Consortium

Rate of Progression of PCDH15-Related Retinal Degeneration in Usher Syndrome 1F (RUSH1F)

Funded by: FoundationFighting Blindnessand Usher 1F Collaborative

Version Number: 1.0

21-Dec-2020

# **Key Roles and Signature Page**

# Rate of Progression of PCDH15-Related Retinal Degeneration in Usher Syndrome 1F (RUSH1F)

Protocol Identifying Number: RUSH1F Version Number: v1.0 21-Dec-2020

| RUSHF Protocol Chair | |
|----------------------------------|---------------------------|
| Name, degree | Katarina Stingl M.D. |
| Signature/Date | |
| JCHR RUSH1F Protocol<br>Director | |
| Name, degree | Allison Ayala, MS |
| Signature/Date | |
| FFB Representative | |
| Name, degree | Todd Durham, PhD |
| Signature/Date | |
| Statistician | |
| Name, degree | Maureen MaguirePhD, FARVO |
| Signature/Date | |

# TABLE OF CONTENTS

| CHAPTER 1: BACKGROUND INFORMATION | 1.5 |
|---------------------------------------------------------------|-----|
| 1.1 Introduction | 15 |
| 1.2 Scientific Rationale for Study Design | 1.7 |
| 1.3 Study Objectives | 17 |
| 1.4 General Considerations | 17 |
| CHAPTER 2: STUDY ENROLLMENT AND SCREENING VISIT | 19 |
| 2.1 Participant Recruitment and Enrollment | |
| 2.1.1 Participant Recruitment Goals and Strategy | 19 |
| 2.2 Informed Consent and Authorization Procedures | 20 |
| 2.3 Screening Visit | 20 |
| 2.3.1 Eligibility Criteria | 21 |
| 2.3.1.1 Participant Criteria | 21 |
| 2.3.1.2 Ocular Criteria | 22 |
| 2.3.2 Screening Data Collection and Testing | 22 |
| 2.3.3 Initial Screen Failures | 23 |
| 2.4 Genetic Screening Phase | 23 |
| 2.4.1Genetic Screen Failures | 25 |
| 2.4.2 Genetics Committee Review | 25 |
| 2.5 Participants Enrolled into the Natural History Study | 25 |
| CHAPTER 3: NATURAL HISTORY STUDY PROCEDURES | 26 |
| 3.1 Baseline Visit | 26 |
| 3.2 Baseline Testing Procedures | 26 |
| 3.3 Follow-up Visits | 27 |
| 3.3.1 Followup Visit Testing Procedures | 28 |
| 3.3.2 Unscheduled Visits | 28 |
| 3.4 Personnel and Equipment Requirements for Study Procedures | 29 |
| CHAPTER 4: UNANTICIPATED PROBLEMS AND ADVERSE EVENT REPORTING | 31 |
| 4.1 Unanticipated Problems | 31 |
| 4.2 Adverse Events | 31 |
| 4.2.1 Definition | 31 |
| 4.2.2 Reportable Adverse Events | 32 |
| 4.2.3 Relationship of Adverse Event to Study Procedure | 32 |
| 4.2.4 Severity (Intensity) of Adverse Event | 32 |
| 4.3 Pregnancy Reporting | 33 |

| CHAPTER 5: MISCELLANEOUS CONSIDERATIONS | 34 |
|---|---|
| 5.1 Treatments During the Study | 34 |
| 5.1.1 Treatment for CDH15Related Retinal Degeneration | 34 |
| 5.1.2 Treatment for Cystoid Macular Edema | 34 |
| 5.1.3 Intraocular Surgical Procedures | 34 |
| 5.2 Risks and Benefits | 3.4 |
| 5.2.1 Risks and Discomforts | 34 |
| 5.2.2 Benefits | 35 |
| 5.3 Collection of Pr∉xisting Conditions and Medications | 35 |
| 5.4 Participant Compensation | 35 |
| 5.5 Participant Withdrawal | 35 |
| 5.6 Confidentiality | 35 |
| CHAPTER 6: STATISTICAL CONSIDERATIONS | 36 |
| 6.1 Sample Size | |
| 6.1.1 Sample Size Considerations for Evaluating Percent Change from Baseline | |
| to 4 Years (All Outcomes) | 36 |
| 6.1.2 Sample Size Considerations for Comparing Percent Change from Baseline | |
| to 4 Years within Subgroups of Interest (All Outcomes) | 37 |
| 6.1.3 Sample Size Considerations for Precision of the Estimate of the Correlation | |
| between Eyes. | |
| 6.1.4 Final Sample Size Justification. | |
| 6.2 Data Analysis | |
| 6.2.1 Primary Objectives Analyses | |
| 6.2.2 Interim Data Analysis | 42 |
| CHAPTER 7: DATA COLLECTION AND MONITORING | 43 |
| 7.1 Case Report Forms and Other Data Collection | 43 |
| 7.2 Study Records Retention | 43 |
| 7.3 Quality Assurance and Monitoring | 43 |
| 7.4 Protocol Deviations. | 44 |
| CHAPTER 8: ETHICS/PROTECTION OF HUMAN PARTICIPANTS | 45 |
| 8.1 Ethical Standard | |
| 8.2 Institutional Review Boards and Ethics Committees | |
| 8.3 Informed Consent Process | |
| 8.3.1 Consent Procedures and Documentation | |
| 8.3.2 Participant and Data Confidentiality. | |
| 8.4 Stored Specimens. | |

# LIST OF ABBREVIATIONS

| ABBREVIATION | DEFINITION |
|---|---|
| ACMG | American College of Medical Genetics |
| ADRP | Autosomal dominant retinitis pigmentosa |
| AE | Adverse Event |
| ANCOVA | Analysis of covariance |
| BCVA | Best corrected visual acuity |
| BRVT | Berkeley Rudimenatry Vision Test |
| CC | Coordinating Center |
| CFR | Code of Federal Regulations |
| CGA | Central Genetics Auditor |
| CI | Confidence interval |
| CME | Cystoid macular edema |
| CSF | Contrast Sensitivity Function |
| DHA | Docosahexaenoic acid |
| EC | Ethics Committee |
| ERG | Electroretinogram |
| ETDRS | Early Treatment of Diabetic Retinopathy Study |
| EVA | Electronic Visual Acuity |
| EZ | Ellipsoid Zone |
| FAF | Fundus Autofluorescence |
| FFB | Foundation Fighting Blindness |
| FST | Full-field stimulusthreshold |
| GCP | Good Clinical Practice |
| ICF | Informed consent form |
| ICH | International Committee of Harmonisation of Technical Requirements for Pharmaceuticals fo Human Use |
| IOP | Intraocular Pessure |
| IRB | Institutional Review Board |
| IS/OS | Inner Segment/ Outer Segment |
| LLVA | Low Luminance Visual Acuity |
| LPV-FVQ II | L.V. PrasaeFunctional Vision Questionnaire |
| MRDQ | Michigan Retinal Degeneration Questionnaire |
| MP | Microperimetry |
| N | Number or sample size |
| OD | Right Eye |
| os | Left Eye |

| ABBREVIATION | DEFINITION |
|--------------|---------------------------------------------------------|
| OU | Both eyes |
| PI | Principal investigator |
| PRO | Patientreported outcomes |
| PROMIS®29 | PatientReported Outcomes Measurement Information System |
| QA | Quality Assurance |
| QC | Quality Control |
| RBM | Risk-Based Monitoring |
| RP | Retinitis pigmentosa |
| SAE | Serious adverse event |
| SD | Standard deviation |
| SD-OCT | Spectral domain opticathoherence tomography |
| SP | Static perimetry |
| TALEN | Transcription activatelike effector nuclease |
| VA | Visual acuity |
| VF | Visual Field |
| VPA | Valproic Acid |

# PROTOCOL SUMMARY

| ITEM | DESCRIPTION |
|---|---|
| Title | Rate of Progression of PCDHRelated RetinaDegeneration in Usher Syndrome (RUSH1F) |
| Précis | This natural history study of patients workCDH15diseasecausing variants will accelerate the development of outcome measures for clinical tensitive, reliable outcome measures of retinal degeneration will greatly facilitate development of treatments for retinitis pigmentosa due CDH15diseasecausing variants. Together these approaches are expected to have an impact on under CDH16 related retinal degeneration, developing experimental treatment protocols, and assessing their effectiveness. |
| | <ol> <li>The goals and expected impact of this natural history study are to: <ol> <li>Describe the natural history of retinal degeneration in patients with lighter diseaseausing variants in the CDH15gene</li> <li>Contribute to the identification expensitive structural and functional outcon measures to use for future multicenter clinical trials@DH15related retinal degeneration</li> </ol> </li> <li>Contribute to the identification of populations for future clinical trials of investigative treatments for CDH15related retinal degeneration</li> </ol> |
| Objectives | <ol> <li>Characterize the natural history of retinal degeneration associated with biallelic diseas@ausing variants in the CDH15gene over 4 years, as measured using functional, structural, and patieported outcome measure</li> <li>Explorewhether structural outcome measures can be validated as surro for functional outcomes in individuals with biallelic diseas@using variants in the PCDH15gene</li> <li>Explore possible risk factors (genotype, phenotype, environmental, and comorbidities) for pogression of the outcome measures at 4 years in individuals with biallelic diseas@ausing variants in the CDH15gene</li> <li>Explore variability and symmetry of left and right eye outcomes over 4 y in individuals with biallelic diseas@ausing variants irhe PCDH15gene</li> </ol> |
| Study Design | Multicenter, longitudinal, prospective natural history study. Participants will be assigned to one of two Vision Cohorts based on visual acuity (VA) and kinetic v fields (VF). |
| Number of Clinical Sites | Approximately 10 |
| Endpoint | <ul> <li>Functional Outcomes:</li> <li>VF sensitivity as measured by static perimetry with quantitative, topographic analysis (Hill of Vision) and assessed by a central reading center</li> <li>Early Treatment of Diabetic Retinopathy Study (ETDRS) Bestected visual acuity (BCVA) letter score as measured on the Electronic Visual Acuity (EV system or ETDRS charts. Berkeley Rudimentary Vision Test (BRVT) will be used for patients unable to see letters</li> <li>Mean retinal sensitivity as measured by funguisdedmicroperimetry (MP) and assessed by a central reading center at selected sites with requisite equipm</li> <li>Full-field retinal sensitivity as measured by ftield stimulus threshold (FST) testing to blue, white and red stimuli</li> </ul> |

| ITEM | DESCRIPTION |
|---|---|
| | <ul> <li>Best corrected low luminance visual acuity (LLVA) letter score</li> <li>Contrast sensitivity function (CSF) as measured by the OSDOE VectorVision chart</li> <li>Structural Outcomes:</li> <li>Ellipsoid zone (EZ) area as measured by spectral domain optical coherence tomography \$D-OCT) and assessed by a central reading center</li> <li>Explore qualitative categorization of Fundus Autofluorescence (FAF) pattern assessed by a central reading center</li> <li>Explore quantitative measures of FAF as assessed by a central reading cer</li> <li>Patient Reported Outcomes (PRO):</li> <li>Adults (18 years or older)</li> <li>Michigan Retinal Degeneration Questionna MRDQ)</li> <li>The MRDQ is a patient reported outcomes instrument for Inherit Retinal Degeneratiowith 59 questions and contains seven domai which are; central vision, color vision, contrast sensitivity, photosensitivity, scotopic function, mesopic and photopic periphological photosensitivity, scotopic function, mesopic and photopic periphological photosensitivity, and activities are pression; anxiety; physical function; pain interference fatigue; sleep disturbance; and ability to participate in social role and activities. The seven domains cover the mostantaveas of self-reported health for most people with chronic illness. There is also one 1-point rating scale for pain intensity.</li> <li>Children (less than 18 years)</li> </ul> |
| | <ul> <li>L. V. PrasaeFunctional Vision Questionnaire (LVPVQ II)</li> <li>The LVP-FVQ-II is a selfreported questionnaire ith 23 questions that will be administered to minor participatos assess selfeported functional vision problems.</li> </ul> |
| Population | <ul> <li>Key Eligibility Criteria: <ul> <li>The entire list of eligibility criteria is in protocol secti@r8.1 and must be reviewed at the Screening Visit. All eligibility criteria must be meteroroll into the genetic screening phase A key subset of those eligibilityriteria includes the following.</li> </ul> </li> <li>Age ≥ 8 years of age <ul> <li>Clinical diagnosis of retinal dystrophy</li> <li>Must meet one of the Genetic Screening Criteria:</li> <li>Screening Group A: At least 2 diseasecausing variants in the PCDH15genewhich arehomozygous or heterozygouis trans, based on report from a clinically certified lator a report from a research lab that has been-approved by the study Genetics Committee)</li> </ul> </li> </ul> |

| ITEM | DESCRIPTION |
|---|---|
| | <ul> <li>Screening Group B: Only 1 diseasecausing variant in the PCDH15gene, basedn a report from a clinically certified lator a report from a research lab which has been preroved by the study Genetics Committee)</li> <li>Screening Group C: At least 2 diseasecausing variants in the PCDH15genewhich areunknown phase based a report from a clinically certified lab(or a report from a research lab which has be pre-approved by the study Genetics Committee)</li> <li>Participants eligible upon initial screening will continue to the genetic screening phase. Following the genetiscreening phase, to be eligible to roll in the study cohort, the following must be documented:</li> <li>Final Study Cohort Criteria: At least 2 diseasecausing variants in the PCDH15genewhich arehomozygous or heterozygouis trans, based on report from a clinicallycertified lab(or a report from a research lab that has been preproved by the study Genetics Committee), condition Auditor (CCA)</li> </ul> |
| Sample Size | Central Genetics Auditor (CGA). Recruitment will be tracked within Vision Cohodefined as follows. Sample size rationale is detailed in protocsection6.1. |
| | <ul> <li>Vision Cohort 1: ~25 participants with the better eyeScreening Visit visual acuity ETDRS letter score of 54 or more [approximate Snellen equivaler 20/80 or betterand visual field diameter 10 degrees or more in every meridian of the central field</li> <li>Vision Cohort 2: ~15 participants with the etter eyeScreening Visit visual acuity ETDRS letter score of 4538 [approximate Snellen equivalent 20/10 20/400]or (visual acuity ETDRS letter score of 54 or more [approximate Snellen equivalent 20/80 or betterid visual field diameter less than 10 degrees in any meridian of the central field)</li> </ul> |
| | The better eyes defined as the eye with better Screening Visit ETDRS VA. I both eyes have the same VA (defined as the same Snellen equivalent), thei determination will be made at investigator discretion as the eye with better fixation or cleaer ocular media topermit highest quality retinal imaging. |
| | The visual field (VF) is defined as a clinically determined kinetic <b>VP</b> e performed within the last 18 months prior to or including the Screening Visit |
| | VF diameter ≥10° in every VF diameter <10° meridian in any meridian 20/80 or better 20/10020/400 Vision Cohort 1 Vision Cohort 2 Vision Cohort 2 Vision Cohort 2 |
| | Initial recruitment goals will be as follows: |

| ITEM | DESCRIPTION |
|---|---|
| | <ul> <li>40 participanteenrolled into the study cohor(tVision Cohorts 1 and 2, combined)</li> </ul> |
| | If recruitment is not at a rate to meet the initial goals, an interim assessment of feasibility may be made by the FFB Consortium Executive Committee inimum of 20 participants enrolled in Vision Cohorts 1 and 2 bimed will be targeted. |
| Participant Duration | From the time of screening until the-#8onth visit: Approximately 51 Months |
| | <ul> <li>ScreeningBaseline Visit (~ 3 months)</li> </ul> |
| | <ul> <li>Baseline Visit– 48-month Followup Visit (~ 48 months)</li> </ul> |
| Protocol<br>Overview/Synopsis | <ol> <li>Investigator reviews patient's current genetic report as meeting one of the Genetic Screening Criterand any other eligibility criteria that can be evaluat based on medical history</li> <li>Consent participant according to overseding itutional Review Board (IRB)/Ethics Committee (EC) requirements</li> <li>Obtain ID on study website tenroll into initial screening</li> </ol> |
| | 4. Complete a Screening Visit to determine eligibility, Visionhort and Genetic Screening Group. Participants meeting criteriactorinue will enroll into the genetic screening phase(See flow chart in next section for details) |
| | <ol> <li>Complete genetic screening according to the requirements for the given Ge<br/>Screening Group. Participants meeting criteria to continue widl into the<br/>study cohort. (See flow chart in next section for details)</li> </ol> |
| | 6. Participants whenroll into the study cohort will return to the clinic within 90 days of the Screening Visit date to start baseline testing, and no late0than daysafter receiving confirmation of meetinginal study cohort criteria from the CGA |
| | 7. All participantswho enroll into the study cohort will return to the clinic at 12, 24, 36 and 48 months from the baseline visit start date for fullpwisits. |
| | 8. After the 48month follow-up visit, participation in thetudywill be completed |

#### 1

# SCHEMATIC OF STUDY DESIGN



2

4 5

6



#### **Genetic Screening Criteria**

One of the following criteria must be met to enter the Genetic Screening Phase:

- <u>Screening Group A:</u> At least 2 disease-causing variants in the gene which are homozygous or heterozygous in trans,
  based on a report from a clinically-certified lab (or a report from a research lab that has been pre-approved by the
  Genetics Committee)
- Screening Group B: Only 1 disease-causing variant in the gene, based on a report from a clinically-certified lab (or a report from a research lab which has been pre-approved by the Genetics Committee)
- <u>Screening Group C</u>: At least 2 disease-causing variants in the gene which are unknown phase, based on a report from a clinically-certified lab (or a report from a research lab which has been pre-approved by the Genetics Committee)

#### Final Study Cohort Criteria

At least 2 disease-causing variants in the gene which are homozygous or heterozygous in trans, based on a report from a clinically certified lab (or a report from a research lab that has been pre-approved by the study Genetics Committee), and confirmed by a Central Genetics Auditor (CGA).

# 

# SCHEDULE OF STUDY VISITS AND PROCEDURES

#### 11 Visit Schedule

| Visit | Screening | Baseline | 12M | 24M | 36M | 48M |
|---|---|---|---|---|---|---|
| Visit Target Windows | (up to Day -90) a | | Wk 52 ± 4° | Wk<br>104± 4° | Wk<br>156±4° | Wk<br>208±4° |
| Participant-Level Procedures | | | | | | |
| Informed Consent | Х | | | | | |
| Demographics/Screening Medical History (including-pxisting | Х | | | | | |
| conditions, patienteported daily activities and medications) | ^ | | | | | |
| Concomitant Medications/Adverse Events | | Х | X | X | Х | Х |
| Patient Reported Outcome (Adults: MRDQ and PROMIS® 29; Children: LPVFVQ II) | | Х | | X | | Х |
| Audiology History | | Х | | | | |
| Pre-cochlear implant audiogram | | Х | | | | |
| Ocular Procedures- All testing performed in each eye | | | | | | |
| Complete Ophthalmic Exam | Х | | Х | Х | Х | Х |
| Visual acuity (including efraction, ETDRS, BRVT if needed, LLVA if needed) | Х | X <sup>h</sup> | Х | Х | Х | Х |
| Contrast Sensitivity(VectorVisionCSV-1000E) | | Х | Х | Х | Х | Х |
| SD-OCT with measurement of EZ area (Heidelberg Spectra | | Х | Х | Х | Х | Х |
| Axial Length and Corneal Curvatureeasurements | | Х | | | | |
| Near Infrared Reflectance Photos (Heidelberg Spectwattis 55degree lens | | Х | | | | |
| Fundus Autofluorescence (Optowhere available | | Х | Х | Х | Х | Х |
| Full-field Stimulus Threshold (Diagnosys Esp)o | | Х | Х | Х | Х | Х |
| Static perimetry (Octopus 900 Pro) | | Χď | Х | Х | Х | Х |
| Fundus guided microperimetry (MAIA) | | Χď | Х | Х | Х | Х |
| Kinetic VF III4e for Vision Cohort definition only | X <sup>f</sup> | | | | | |

- a. All Screening Visit testing must be completed on the same day
- b. Baseline Visit date (defined as the start date of all Baseline testing) must latter than 80 days after receiving confirmation of meeting in all study cohort criteria from the CGA (and possible, within 90 days of the Screening Visit date). All Baseline testing hould be completed within 7 days of the Baseline Visit date PROs as specified.
- c. All Follow up visit testing must be completed on the same elagept PROs as specified.
- d. For static perimetry and microperimetry, all Vision Cohort 1 and 2 participants will complete two **teasts** late The results will be compared according to **this** ual field criteria to determine if a third test is needed.
- e. Ophthalmic exam includes slitmp biomicroscopy, indirect ophthalmoscopy and intraocular pressure (IOP). IOP measurements will be taken prior to pupil dilation will take place at approximately the same time of the day at each visit and with the same quipment
- f. Kinetic VF III4e performed within the last 18 months prior to or including the Screening Visit date for Vision Cohort determination only
- g. May be completed in person or remotely any time within the sallowable window of the associated visit window (not required to be the same day as the rest of the visit).
- h. If the Baseline visit date is more than 90 days after the Screening Visit date, all Visual acuity procedures must also be completed
- i. Required for all sites exce**pt**ith the exception of any site with equivalent equipment approved by the reading center and operations committee

33

# Chapter 1: Background Information

1.1 Introduction

Usher syndrome (USH), is a neurosensory distractempacts ision and learing, inherited in an autosomal recessive way. It is characterized by the combination of hearing impairment up to deafness and retinal dystrophy (retinitis pigmentosa, & Pa) some cases vestibular and olfactory deficits. The three main clinical subtypes sown are USH1, USH2 and USH3. USH type 1 (USH1) patients are born completely detained patients experience other polications such as delayeds itting and walking age due to vestibular proble Rewith night blindness typically diagnosed by 10 years of age. In USH2 patients, hearing impairment is less pronounced and the patients do not experience lance deficit. In most cases, this subtype so not progress over time. Night blindness normally occurs later than in 9518143 account for 2% of patients and found mostly in Finland and Ashkenazi. Jewis type the hearing impairment is progressive, and a balance defect may be pfesent

USH1F is a subtype of USH1 caused by albelic mutations of the USH1F gene, also called protocadherin 15 (PCDH15). This gene has been localized in ear hair cell stereocilia and outer segments of primates' retinal photoreceptors; strongPCDH15 activity has been described in cones, but also diffusely in rods through the whole photoreceptor all the remajority of PCDH15 mutations leading to USH1F are localized in the ectodomains of the protein, but not in the transmembrane domain or the cytoplasmic domain, the latter two being probably important outside of the hearing and visual system. It is result that PCDH15 might have a role in the morphogenesis and cohesion of stereocilia bundles and retinal photoreceptor cell maintenance or function Protocadherin 15 deficiency leads to functionally impaired cones and rods with abnormally shaped outer segression.

PCDH15 has been linked to congenital deafness or its syndromic form USAMBitionally, digenic inheritance of Usher syndrome USH1D/F has been described in patients with heterozygous mutations in both CDH23 arcale DH15 genes The prevalence of USH1 is around 1-9/100,000; the prevalence of USH1F is not precisely with due to its rarity but might be around 10 % of all USH1 patients

The current knowledge about the naturalree of USH1F is limited, as resystematic observational trials of the retinal phenotype vebeen published. The phenotype and fast time course of the retinal degeneration in USHIS comparable with the phenotype of USH1 in general, which is characterized by profound pre-lingual deafness, vestibular ataxia, and childhood onset of retinitis pigmento 12 at 2

A large cohort of 268 USH patients in a multicement uropean tsudy TREATRUSH (https://cordis.europa.eu/project/rcn/95259\_en.htmals) conducted tonderstand the genotype phenotype correlations of USthidenabled some insight into the subgroups of phenotypes of USH1. The analysesom this study indicated and visual fields and visual acuity as function of the patients' age corresponds to the changes of the USH1 cohort in general. 12

Hearing loss is treatable with cochlear implants in many patients with U\$\textit{HoWe}\text{ever,the} therapy for treating the retinal phenotype is still in preclinical research. Gene replacement

therapy, similar as the first approved AAV (adeno associated virus) mediated subretinal gene therapy for RPE65 retinitis pigmentosa, is not possible in USHIERo the large size of the PCDH15 gene.

Genebased therapies such as dwattors, gene editing or mini geness, dsuppression of several PCDH15 mutations by aminoglycosidese have nexamined. Aminoglycosides can influence the translation of mRNA improtein by inhibiting ribosomal proofreading, thus, leading to readhrough of nonsense mutations partial readthrough of PCDH15 nonsense mutations leading to various levels of the fleshight proteinwas shown by aminoglycosides in vitro and ex vivo<sup>13</sup> However, more preclinical and clinical research is needed to whether these approaches an restore vision in patients with USH16F slowdown the degeneration process leading to blindness.

The clinical research in therapy trials for other types of syndromic mosyndromic RP shows that valid readouts are one of the most important aspects of clinical trials. Morphological readouts have improved with high resolution retinal imaging such as spectral domain OCT (SD OCT) and became standard in clinical follows and clinical trials due to its objectivity and lower variability than psychophysical functional tests

For functional tests of the retinasychophysical examinations of visual fields and best corrected visual acuity (BCVA) as well as contrast vision (or low luminance BCVA) are commonly used but describing only foxed cone vision. Further, fundus guided mesopic microperimetry has been used widely in clinical trials of inherited retinal degenerations. However, due to the mesopic range of the stimuli, the method is not sensitive enough to testsiod. Additionally, in retinal degeneration with increasing dandapted rod thresholds, the mesopic testing is not able to distinguish between the degenerating rod system and the healthy or degenerating cone system.

With respect to the knowledge of the progrie of the cone and rod degeneration and future therapy approaches, a clear differentiation of the rod and cone function is desirable. Routinely used objective readouts of the photoreceptors such as scotopic and photopic extends phy (ERG) are usally non-recordable already in early stages of the retinal degeneration, including RP in USH1 patient. Therefore, the fulfield ERG is not apractical follow-up readout for the natural course dust or therapy interventions. A psychophysical test of the delatated thresholds, FST (fulfield stimulus threshold) with chromatic stimuli is better suited to describe the deterioration of the retinal progriess even in late stages of RP18

Although these scotopic readouts are widely used, they do not possess the ability to show the local retinotopy of the rod system. A method who was evaluate the local rod function is dark adapted chromatic perimetry (DAC). This method has also earlier been applied in patients with RP.<sup>19,20</sup>A novel, shortened protocol for application in RP trials has been proposed recently with duration of around 7 minutes, intervisit repeatability of 7.6  $\pm$  2.8 dB for cyan and 5.9  $\pm$  1.7 dB for red stimuli and ability to detect the dal rod rescue after gene ther application application and 1.2 dB.

Further, novel diagnostic development has been introduced, enablinger tive, retinotopically correct evaluation of the rod and cone system by analyzing the pupil response to local stimuli<sup>23</sup> The chromatic pupil campimetry, although not broadly available, is a tool for

- evaluation of the function of both photoreceptors separately be bjective way, with a superior intervisit repeatability compared to DAC
- 127

142

143

144

145

146

147

149

150

151

152

153

154

155

156 157

158

159

- 128 In respect to the promising therapy approves in RP, including the retinal phenotypes of USH1,
- 129 clinically acceptable tests of the local rod and cone function, supporting the morphological
- 130 evaluations such as OCT are needed. Only understanding the dynamic of the cone and rod
- degeneration over tienin a retinotopically correct manner can enable us to understand the
- 132 natural history of the disease and to evaluate eventual therapy safety and efficacy in the future
- 133 1.2 Scientific Rationale for Study Design
- 134 A prospective natural history studythe gold standard for tracking the course of disease. The
- 135 knowledge of the course patients with PCDH15 mutations will guide the planning of future
- 136 controlled treatment trialsdentifying the most snsitive and reliable outcome measures of
- retinal degeneration wigreatly facilitate development of treatments maximum efficiency
- 138 Together these approaches are expected to have an impact on unders Parability 5 related
- retinal degeneration, developing/estigational reatment protocols, and assessing in
- 140 effectiveness.
- 141 The goals and expected impact of this natural history study are to:
  - Describe the natural history of retinal degeneration in patients with biallelic mutations in the PCDH15gene
  - Contribute to the identification exensitive structural functional outcome measures to use for future multicenter clinical trials PCDH15 related retinal degeneration
  - Contribute to the identification of opulations for future clinical trials of investigative treatments foPCDH15related retinal degenerate

#### 148 1.3 Study Objectives

- 1. Characterize the natural history of retinal degeneration associated with biallelic pathogenic mutations in the CDH15gene over 4 years, as measured using functional, structural, and patient ported outcome measures
- 2. Explorewhether structural outcome measures can be validated as surrogates for functional outcomes in individuals with biallelic pathogenic mutations in POPH15 gene
- 3. Explorepossible risk factors (genotype, phenotype, environmental, and comorbidities) for progression of the outcome measures at 4 years in individuals with biallelic pathogenic mutations in the CDH15gene
- 4. Explore variability and symmetry of left and right eye outcomes over 4 years in individuals with biallelic pathogenic mutations in the PCDH15 gene
- 160 1.4 General Considerations
- 161 The study is being conducted in compliance with the ethical principles that have their origin in
- the Declaration of Helski, with the protocol described herein, and with the standards of Good
- 163 Clinical Practice (GCP)Employing a prospective longitudinal study design is advantageous
- because it reflects systematic method of data collection study design incorporates several
- 165 strategies to minimizbias detailed belowusing consideration from "RareDiseases: Natural

| 166<br>167<br>168<br>169 | History Studies for Drug Development: Guidance for Industry, Draft Guidandeneseare considered standard for treatment trials and will enhance the translation of the data from this study to a treatment trial. |
|---|---|
| 170<br>171 | • Establishing standardized testing procedures and specific required equipmatent investigators, leading to greater consistency and precision in the information explication. |
| 172 | <ul> <li>Training and ertification of study staff who will perform following procedures</li></ul> |
| 173 | related to the primary outcom &P, OCT, MP, FAF) by a Reading Center. The Reading |
| 174 | Center will grade test results a uniform manner independently from study sites |
| 175 | <ul> <li>Use ofstandard, consistent definitions pre-existing medical conditions, medications</li></ul> |
| 176 | and treatment and adverse event (AEs) across all clinical sites |
| 177 | <ul> <li>A consistent schedule of followp visits for all participants whitestablished visit time</li></ul> |
| 178 | frames |
| 179 | <ul> <li>A coordinating cente(CC) is responsible for monitoring the conduct of the study to</li></ul> |
| 180 | ensure adherence to protocol |

# Chapter 2: Study Enrollment and ScreeningVisit

- 182 2.1 Participant Recruitment and Enrollment
- 183 Study participants will be recruited from proximately 10 clinical sites worldwide. All eligible
- participants will be included without regard to gender, race, or ethrential eligibility will
- be assessed during a routine examination by an inatestigrior to obtaining informed consent,
- as part of usual carthrough referrals from other providersself-referral

#### 2.1.1 Participant Recruitment Goals and Strategy

Recruitmentwill be tracked withintwo Vision Cohorts defined as follows Sample size rationale is detailed in insection 6.1.

- Vision Cohort 1: ~25 participants with the *better eye* Screening Visit visual acuity ETDRS letter score of 54 or more [approximate Snellen equivalent 20/80 or better] and visual field diameter 10 degrees or more in every meridian of the central field
- Vision Cohort 2: ~15 participants with the *better eye* Screening Visit visual acuity ETDRS letter score of 19-53 [approximate Snellen equivalent 20/100 20/400] <u>or</u> (visual acuity ETDRS letter score of 54 or more [approximate Snellen equivalent 20/80 or better] <u>and</u> *visual field* diameter less than 10 degrees in any meridian of the central field)

The better eyes defined as the eye with better Screening Visit ETDAS If both eyes have the same A (defined as the same Snellen equivalent), then the determination we made at investigator discretion as the eye with better fixation or clearly are media to permit highest quality retinal imaging.

The visual field (VF) is defined as the clinically termined kinetic/F III4e performed within the last 18 months prior to or including the reening Visit date.

VF diameter VF diameter ≥10° in every control version veridian veridian

20/80 or better 20/10020/400

Vision Cohort 1 Vision Cohort 2 Vision Cohort 2 Vision Cohort 2

188

189

190 191

181

187

The Foundation Fighting Blindness (FFB) nsortium Executive Committee will review recruitment progress and feasibility at regular intervaliatial recruitment goalswill be as follows:

- 40 participantsenrolled into the studycohort (Cohorts 1 and 2 combined)
  - If recruitment is not at a rate to meet the initial goals, an interim assessment of feasibility maybe made by the FFBonsortiumExecutive CommitteeA minimum of 20 participants enrolled inVision Cohort1 and VisionCohort2 combinedwill be targeted

194 195 196

- 197 Participants will not be counted as a senrolled into the study cohort until initial screening and
- 198 genetic screening haveenconfirmed as a successsections 2.3 and 2.4). This means that
- more participants will be screened than noted above the number and reasons for screen failures
- 200 will be tracked. It is also possible that some participants will have completed & eening Visit
- and and an another and a second a second and a second
- 202 above therefore the final enrolled numbers may be larged.limit over-enrollment clinical
- sites will be notified as the recruitment goals near completion, efforts with ade to accurately
- 204 predictnumbers in the genetic screening queund consent and creening f participants which
- 205 could contribute to ver-enrollmentin a given Vision Cohortmay be paused
- 206 2.2 Informed Consent and Authorization Procedures
- 207 Potential eligibility may be assessed as part of a routine examination an investigator prior
- 208 to obtaining informed consent, as part of usual, day referral from another physician self-
- 209 referral Before completing any procedures or collecting any data that are not part of usual care,
- 210 written informed consent will be obtained sing consent documentation approved by the
- 211 overseeing IRB/ E.
- 212 The study protocol will be discussed with the potential studio protocol will be discussed with the protocol will be discussed with the protocol will be discussed with the protocol will be
- 213 potential study participant will be given the Informed Consent (100m) to read. Potential
- 214 study participants with severe vision impairment rhay presented with a Short Forton be read
- 215 aloud by a clinical staff memberthey preferfollowing the overseeing IRB/Œrequirements.
- 216 Potential study participants will be encouraged to discuss the study with family members and
- 217 their personal physicians(s) before deciding whether to participate in the study.
- 218 As part of the informed consent process, each participant will be asked to sign an authorization
- 219 for release of personal information. The investigator, or his or her designee, will review the
- 220 study-specific information that will be collected and to whom that information beild is closed.
- 221 After speaking with the participant, questions will be answered about the details regarding
- 222 authorization.
- 223 A participant is considered into the initial screening when the CF has been signed
- and a participant ID has been obtained the study website.
- 225 An immediate family members) of studyparticipants may be asked to articipate infamily
- membergenetic testing as part of the genetic screening phastenese cases, family members)
- will be asked to provide a saliva samples (critical in section 2.4). An electronic consent form
- 228 will be reviewed and signed the family member(s) in order to obtain permisstorcollect a
- 229 saliva sample.
- 230 2.3 Screening Visit
- 231 After the ICF has been signed potential participant will bevaluated for study eligibility
- through the elicitation of a medical history, performance of ophthalmic tests as described below,
- and genetic testing applicable. The Screening Visit date will be the date the Screening Visit
- 234 testing procedures starte All Screening Visit testing procedures il be complete on this date.

| 235 | 2.3.1Eligibility Criteria |
|---|---|
| 236<br>237 | To be eligible to <b>enroll into the genetic screening phase,</b> a study participant must meet all the inclusion criteria and none of the exclusion criteria at the Screening Visit. |
| 238 | 2.3.1.1 Participant Criteria |
| 239 | Participant Inclusion Criteria |
| 240<br>241 | Participantsmust meetall the following inclusion criteria at the Screening Visitin orderto be eligible to enroll into the genetic screening phase |
| 242<br>243<br>244<br>245<br>246<br>247<br>248<br>249<br>250<br>251<br>252<br>253<br>254<br>255<br>256<br>257<br>258 | <ol> <li>Willing to participate in the study and able to communicate consent during the consent process</li> <li>Ability to return for all study visits over 48 months</li> <li>Age ≥ 8 years</li> <li>Not planning to enroll in an experimental clinical trial for the treatment of PCDH15 for the duration of this study</li> <li>Must meet one of the Genetic Screening Criteria, defined below: <ul> <li>Screening Group A: At least 2 diseasecausing variantsin the PCDH15gene which arehomozygousor heterozygousin trans, based on report from a clinically certified lab (or a report from a research lab that has beerappeoved by the Genetics Committée)</li> <li>Screening Group B: Only 1 diseasecausing variantin the PCDH15 gene, basecon a report from a clinically certified lab (or a report from a research lab which has been prapproved by the enetics Committée)</li> <li>Screening Group C: At least 2 diseasecausing variants in the PCDH15 gene which areunknown phase basecon a report from a clinically certified lab (or a report from a research lab which has beenapperoved by the enetics Committee)</li> </ul> </li> </ol> |
| 260<br>261<br>262<br>263 | <b>Note pertaining to all Screening Groups:</b> if a participant has a variant(s) of unknown significance, he/she would still qualify if there is at least 1 disease-causing variant(s) on the PCDH15 gene. <b>Participant Exclusion Criteria</b> |
| 264<br>265 | Participantsmust not meeting of the following exclusion criteria at the Screening Virsitrder to beeligible to enroll into the genetic screening phase |
| 266<br>267<br>268<br>269<br>270<br>271<br>272<br>273 | <ol> <li>Mutations in genes that cause autosomal dominant retinitis pigmentosa (ADRP), X-linked retinitis pigmentosa (RP), or presence of biallelic mutations in autosomal recessive RP/retinal dystrophy genes other than PCDH15</li> <li>Expected to enter experimental treatment trial at any time during this study</li> <li>History of more than 1 year of cumulative treatment, at any time, with an agent associated with pigmentary retinopathy (including hydroxychloroquine, chloroquine, thioridazine, and deferoxamine)</li> </ol> |
| 274 | <b>Note:</b> Pregnant women are not being specifically excluded from participation. |

| 276 | 2.3.1.2Ocular Criteria |
|---|---|
| 277<br>278<br>279 | Ocular Inclusion Criteria Both eyes mst meetall the followingat the Screening Visfor a participanto be eligible to enroll into the genetic screening phase |
| 280<br>281<br>282<br>283 | <ol> <li>Clinical diagnosis of retinal dystrophy</li> <li>Clear ocular media and adequate pupil dilation to permit good quality photographic imaging</li> </ol> |
| 284<br>285<br>286 | Ocular Exclusion Criteria If either eye has any of the following the Screening Vişitheparticipantis not eligibleto enroll into the genetic screening phase |
| 287<br>288<br>289<br>290<br>291<br>292<br>293<br>294<br>295<br>296<br>297<br>298<br>299<br>300<br>301<br>302<br>303<br>304<br>305<br>306<br>307<br>308<br>309 | <ol> <li>Current vitreous hemorrhage</li> <li>Current or any history of tractional or rhegmatogenous retinal detachment</li> <li>Current or any history of (e.g., prior to cataract or refractive surgery) spherical equivalent of the refractive error worse than -8 Diopters of myopia</li> <li>History of intraocular surgery (e.g., cataract surgery, vitrectomy, penetrating keratoplasty, or LASIK) within the last 3 months</li> <li>Current or any history of confirmed diagnosis of glaucoma (e.g., based on glaucomatous VF changes or nerve changes, or history of glaucoma filtering surgery)</li> <li>Current or any history of retinal vascular occlusion or proliferative diabetic retinopathy</li> <li>History or current evidence of ocular disease that, in the opinion of the investigator, may confound assessment of visual function</li> <li>History or evidence of active treatment for retinitis pigmentosa that could affect the progression of retinal degeneration, including: <ul> <li>Any use of ocular stem cell or gene therapy</li> </ul> </li> <li>Any treatment withocriplasmin</li> <li>Treatment with an ophthalmic oligonucleotide within the last 9 months (last treatment date is less than 9 months prior to Screening Visit date)</li> <li>Treatment with any other product within five times the expected half-life of the product (time from last treatment date to Screening Visit date is at least 5 times the half-life of the given product)</li> <li>Treatment with Ozurdex (dexamethasone), Iluvien or Yutiq (fluocinolone acctonide) intravitreal implant</li> </ol> |
| 310 | 2.3.2ScreeningData Collection and Testing |
| 311<br>312<br>313<br>314<br>315 | The study design schematic at the beginning of the protocol shows the flow of the Screening Visit. The following procedures will be performed at the protocol shows the flow of the Screening Visit. The testing procedures are detailed in the RUSH1FC linical Site Manual of Procedure of the equipment and technician requirements for all testing is section 3.4. All ocular testing will be performed in each eye right eye (OD) first and then left eye (OS). |
| 316<br>317<br>318 | Participants meeting criteria to continue will enerolled into the genetic screening hase (section 2.4. Otherwise the participant will be an initial screen failure (section 2.3.3) The below information will be collected the Screening Visit: |

- 1. Contact information (retained at tblinical site and notentered the study database)
- 2. Inclusion and exclusion criteria assess t(criteria insections 2.3.1.1 and 2.3.1.2
- 3. Demographicsin cluding sex, raceethnicity)

325

326

327 328

329

330

331

332

333

334

335336

337

338

339

340 341

342

343 344

- 4. A medicalhistory will be elicited from the study participant and extraction available medical records, including atient reported daily activities pre-existing medical conditions and medical records.
  - Complete ophthalmic exam. Exam will include stimp biomicroscpy, indirect ophthalmoscopy, and intraocular pressure (IOP). IOP measurements will be taken prior to pupil dilation
    - Genetic screening assessmemulations number and phase of mutations in Production gene, history of consanguinity and collection of theorem genetic report(s) available at the clinical site
      - This includes an assessment that the participant meets three definetic Screening Criteria described in section 2.3.1.1 If the participant does not meet the criteria for one of the Genetic Screening Groups, then theremainder of procedures antesting arenot required. Participantial be discontinued as an initial screen failure per section 2.3.3
  - Visual acuity(including refraction, ETDRS, BRVT if needed, LLVA if needed)
    - > The VA letter score will determine whether LLVA or BRWill be performed. The criteria are defined in the USH1FClinical SiteManual of Proceduse
    - 8. Kinetic VF III4e (or historical measuremeperformed within the last 18 months prior to or including the Screeing Visit date Vision Cohortdetermination based oneye with bettervisual acuity and kinetily F above (criteria insection 2.1.1)
      - ➤ If the participant's determined/ision Cohortis closed for enrollmenthe remainder of procedures and testingenot required. Participantill be discontinueds an initial screen failure per section 2.3.3
      - 2.3.3Initial Screen Failures
- Participants who do nonteetcriteria to continue as notembove will be discontinued as an initial screen failure. The Screening Visit Form will still be completed, entering "Not Done" for testing notinished A Final Status Form will be completed, and the reason for screen failure will be noted.
- 350 2.4 Genetic Screening Phase
- Participants passing the initial screening and enrolling int Genetic Screening Phasewill
- 352 complete the following genetic testing and/or review procedures ording to their Screening
- 353 Group (defined in section 2.3.1.) The study design schematic betbeginning of the protocol
- 354 also summarizethe flow of the Genetic ScreeninghaseMore detailed procedureare specified
- 355 in the RUSH1FClinical Site Manual oProcedures
- All genetic reports noted below to be uploaded to the study website by that stite or Central Lab may be available to and reviewed by α6 eassociated clinicalite, Central

Lab, CGA, Genetics Committee, and investigators involved in oversight of the study (which include the study chair, Operations Committee, Fartal Consortium Executive Committee). All reports will be diglentified prior to uploading

#### Screening Group A

- The clinicalsite will upload supporting genetic documentation (including genetic reports) onto the study website
- A CGA will review thegeneticdocumentation provided by the clinicastite to verify the
  genetic screening at a entry and ppropriated ocumentation of the final study cohort
  criteria (section 2.5) of at least 2 disease ausing variants in the PCDH15 genewhich
  arehomozygous or heterozygous trans. Additional documentation may be requested
  as needed to verify then al study cohort criteria and all genetic screening assessments
  - If final study cohort criteria areverified, participant will be considerent rolled into the study cohort
  - Otherwisetheparticipantwill be agenetic screen failure(section 2.4l)

#### Screening Group Bor C

- The clinical site willupload supporting genetic documentation (including genetic reports) onto the study website
- Participants will be asked to provide a saliva sample, and apparbactst1 first-degree relative to provide a saliva sample for additional gertesting. The first-degree relative(s) will be provided with information on how to provide informed consent and how to complete the saliva kit.
- The participant's and first degree relative(s)'s samples will be shipped to and analyzed by the Central Lab to conduct retinal dystrophypanel genetic testing and termine the presence and number of diseasesing variants on the CDH15gene (Screening Group B only), and the phase of the alleless on the family member testing Groups B and C) The Central Lab will provide these assessments attackenetic repo(ts), which will be uploaded to the study website
  - o If the Central Lab determines there are at least 2 diseas@ausing variants in the PCDH15 genewhich are homozygous or heterozygous rans, the participant's reports will move forward o CGA review
  - Otherwisethe participantwill be agenetic screen failure(section 2.41)
- A CGA will review the reports provided by the clinical saited the Central Lato verify the genetic screening data entry appropriatedocumentation of the study cohort criteria (section 2.5) of at least 2 disease causing variants in the PCDH15 genewhich are homozygous or heterozygous trans. Additional documentation may be requested as needed to verify the all study cohort criteria and all genetic screening assessments
  - If final study cohort criteria areverified, the participant will be considered enrolled into the study cohort
  - Otherwisethe participantwill be agenetic screen failure(section 2.41)

| 397 | 2.4.1GeneticScreen Failures |
|---|---|
| 398<br>399<br>400 | Participants who do not meet criteria to continue as noted above will be discontinued as a genetic screen failure. A Final Status Form will be completed, and the reason for screen failure will be noted. |
| 401 | 2.4.2Genetics Committee Review |
| 402<br>403<br>404<br>405<br>406<br>407 | A Genetics Committervill review the genetic documentation participants with verified final study cohort criteria and enrolled into the study cohort for interpretation evaluation whether the PCDH15 mutations are causative of the iseas (i.e., pathogeni, dikely pathogeni). Details of the process are described in tree SH1FM onitoring Plan Cases that are confirmed as disease causing will remain in the study and will not be considered ineligible, however their data may be analyzed separately from those with pathogenic mutations. |
| 408 | 2.5 Participants Enrolled into the Natural History Study |
| 409<br>410<br>411 | All participantsmeeting initial screening and eligibility criteria (sect206.1) who complete the Genetic Screening Phase (sect204) and meet the final study cohort criteria (defined below) will be considered into the study cohortand will complete the natural history study. |
| 412<br>413<br>414<br>415 | Final Study Cohort Criteria: At least 2 diseasecausing variants in the PCDH15gene which are homozygous or heterozygous trans, based on report from a clinically certified lab (or a report from a research lab that has been appreciated by the study genetics committee), and firmed by aCGA |

| 416 | | | Chapter 3: Natural History Study Procedures |
|---|---|---|---|
| 417 | 3.1 Ba | aseline | Visit |
| 418<br>419<br>420<br>421<br>422<br>423 | Participants meeting criteria to enter the natural history study (section 2.5) will return for a Baseline Visit date within thirty (30) days after receiving confirmation of meeting <b>final study cohort criteria</b> from the CGA. The Baseline Visit date will be documented as the date testing procedures began. All Baseline Visit testing procedures will be completed within seven (7) days of the Baseline Visit date, except PROs as specified below. | | |
| 424<br>425<br>426<br>427<br>428 | for the Baacuity | e studya<br>seline<br>testing | rocedures that apperformed at the Screening Visit willerve as baseline measures and will not be completed again at the Baseline Vīstie only exceptionwill be if Visit date is more thannety (90) days after the Screening Visit date The visual g willneed to be repeated (including refraction, ETDRS, LLWAneeded BRVT if baseline visit is completed more thannety (90) days from the screening visit |
| 429 | 3.2 Ba | aseline | Testing Procedures |
| 430<br>431<br>432<br>433 | detaile<br>and c | edin the<br>ertificat | gprocedureswill be performed the Baseline Visit The testing procedures are eRUSH1FClinical Site Manual of Procedures overview of the equipment tion requirements for all testing is insection 3.4. All ocular testing will be eacheye OD first and the OS. |
| 434<br>435 | 1. | | cal updates, including new/changed adverse events, ocular proç <b>add</b> res cations |
| 436 | 2. | Audio | logy history |
| 437<br>438<br>439<br>440 | | a. | Participantreported audiology history will be collected on the Audi <b>globi</b> story Information Form. This includes history of hearing loss, newborn screening hearing, hearing aid use, cochlear implant use, history of ear infections, history of ear surgery and balance disorders. |
| 441 | 3. | Audio | gram (request the most recent-poæhlear inplant audiogram) |
| 442<br>443<br>444<br>445<br>446 | | a. | The most recentival ableaudiogram prior to cochlear implantial be collected on each participant cluding air conduction threshold and bone conduction threshold The Audiogram Results Form will be completed using the most recent audiogram. The historical audiogram will be sent to the atral study adiologist reviewer, to confirm correct interpretation for the Results Form |
| 447 | 4. | Patier | nt Reported OutcoméAdults: MRDQ and PROMIS®9; Children: LPVFVQ II) |
| 448<br>449<br>450 | | a. | The PROs may be completed in personnemotely (phone or other remote methods) any time within 6 months of the Baseline Visit (not required to be the same day as the rest of the Baseline Visit) |
| 451 | 5. | Contra | astsensitivity |
| 452 | 6. | SD-O | СТ |
| 453 | 7. | Axial | Lengthand Corneal Curvature measurements |
| 151 | Ω | Maarl | nfraredReflectanc&hotos |

| 455 | 9. Full-field Stimulus Threshold |
|---|---|
| 456 | 10. Fundus Autofluorescence (on Optos, where available) |
| 457 | 11. Static perimetry |
| 458<br>459 | <ul> <li>a. Two tests will be performed. The inical sitewill compare the certified technician determined mean sensitivity from test 1 versus test 2</li> </ul> |
| 460<br>461<br>462 | <ul> <li>If the absolute value of the difference betweentwheetests is ≤ 2.4 dB, then<br/>the participant passes static perimetry reliability criteriaæthdrd test isnot<br/>needed</li> </ul> |
| 463<br>464<br>465 | <ul> <li>If the absolute value of the difference betweentwhetests &gt; 2.4 dB then<br/>the participant does not pass static perimetry reliability criteria, and a third<br/>is needed</li> </ul> |
| 466 | 12. Fundusguided microperimetry |
| 467<br>468 | <ul> <li>a. Two tests will be performed. The inical sitewill compare the certified technician determined mean sensitivity from test 1 versus test 2</li> </ul> |
| 469<br>470<br>471<br>472 | <ul> <li>If the absolute value of the difference betweentwhoetests divided by the<br/>average between theim ≤ 50% OR the absolute value of the difference<br/>between the two tests ±s0.5 dB, then the participant passes microperimetry<br/>reliability criteria and third test is not needed</li> </ul> |
| 473<br>474<br>475<br>476 | o If the absolute value of the difference betweentwhetestsdivided by the<br>average between theirs> 50% AND the absolute value of the difference<br>between the two tests is0-5 dB, thenthe participant does not pass<br>microperimetry reliability criteria and third test is needed |

#### 3.3 Follow-up Visits

The Baseline Visit date is considered study day 0, from which follow-up visit windows are timed. The Follow-up Visit date will be the date the Follow-up Visit testing procedures started. All Follow-up Visit testing procedures will be completed on the same date other than the PROs required at the 24 Month and 48 Month Visits, which can be completed  $\pm$  6 weeks of the visits.

Follow up visits will be conducted at:

| Visit | Target | Target Window | Allowable Window |
|----------------|-----------|---------------|------------------|
| 12 Month Visit | 52 Weeks | ± 4 Weeks | ± 6 Weeks |
| 24 Month Visit | 104 Weeks | ± 4 Weeks | ± 6 Weeks |
| 36 Month Visit | 156 Weeks | ± 4 Weeks | ± 6 Weeks |
| 48 Month Visit | 208 Weeks | ± 4 Weeks | ± 6 Weeks |

484 485

486

477

478

479

480 481

482 483

> Visits will be scheduled in the target window. If circumstances do not permit this, visits may be scheduledo extend out to allowable window without being considered a protocol deviation

a thtird tes

| 487<br>488<br>489<br>490 | The reason for scheduling outside the target windownust be documented on the visit form. Visits that occurout of the allowable windowill be used for analysibut will be documented as protocol deviations Details regarding when to consider a visit missed are specified in the RUSH1FC linical Site Manual of Procedures | |
|---|---|---|
| 491 | 3.3.1Follow-up Visit Testing Procedures | |
| 492<br>493<br>494<br>495<br>496 | The following procedures will be performed at freelow-up Visits as noted below The testing procedures are detailed in tReSH1FClinical Site Manual of Procedures noverview of the equipment and certification requirements for all testing securion 3.4. All ocular testing will be performed in acheye OD first and ther OS. | |
| 497<br>498 | | ollowing will be performed athe 12 Month, 24 Month, 36 Month, and 48 Month \sisi s otherwise noted. |
| 499 | 1. | Medical updates, including new/chang@sas, ocular procedures, and medications |
| 500<br>501 | 2. | Patient Reported Outcomes24Month and 48Month visits only(Adults: MRDQ and PROMIS®29; Children: LPVFVQ II) |
| 502<br>503<br>504 | | a. The PROs may be completed in person or remotely (phone or other remote methods) any time within the Allowable Window of the associated visit, (not required to be the same day as the rest of the Follow up Visit). |
| 505<br>506<br>507 | 3. | Complete ophthalmic exam. Exam will include slit-lamp biomicroscopy, indirect ophthalmoscopy, and intraocular pressure (IOP). IOP measurements will be taken prior to pupil dilation |
| 508 | 4. | Visual acuity(including refraction, ETDRSPRVT if neededLLVA if needed) |
| 509<br>510<br>511 | | <ul> <li>a. The visual acuity letter score will determine whether LLVA or BRMT be<br/>performed. The criteria are defined in the SH1FClinical Site Manual of<br/>Procedures</li> </ul> |
| 512 | 5. | Contrast sensitivity |
| 513 | 6. | SD-OCT |
| 514 | 7. | Full-field Stimulus Threshold |
| 515 | 8. | Fundus Autofluorescence (on Optos, where available) |
| 516 | 9. | Static perimetry |
| 517 | 10 | . FundusguidedMicroperimet <b>y</b> |
| 518 | | 3.3.2Unscheduled Visits |
| 519<br>520<br>521<br>522<br>523 | Testing procedures at scheduled is its areat investigator discretion. However, it is recommended that procedures performed ingthese visits follow the standard protocol for each procedure and performed certified personne Unscheduled visits will be recorded the FFBC onsortium study webste. Study images taken during unscheduled visits not require submission to the study website. | |

- 3.4 Personnel and Equipment Requirements for Study Procedures
- The testing procedures are detailed in RNASH1FClinical Site Manual of Procedures overview of the equipment and certification requirements for all testine gas follows.

| Study Procedures | Equipment Required (if applicable) | Who can Perform |
|---|---|---|
| Investigator takingverall responsibility for avisit oversees that consent process was formed in accordance with IB/EC requirements igns off on all eCRFs for a participant, eCRF edits, and protocol deviations | N/A | Certified investigator |
| Coordinator taking responsibility for the visit oversees the data entry aspect of the visit, addresses protocol queries and signs off on deviations | N/A | Certified coordinator |
| Informed consent: explanation/review of study with th potential participanand/or signature of ICF | N/A | Certified investigatocoordinator as permitted by the IREC |
| Signature of Informed Consent Form | N/A | Certified investigator/coordinator as permitted by tht RB/EC |
| Data entry on study website | Computer and internet connection | Certified coordinator<br>(or certified investigator with<br>additional study website<br>certification) |
| Sample collection and shipping | Study will provide necessary<br>materials- detailed in<br>RUSH1FClinical Site<br>Manual of Proceduse | Certified coordinator |
| Collect information regarding medicalhistory, demographics adverse events, medications | N/A | Certified investigator/coordinator |
| Patient Reported Outcomes | Study will provide necessary<br>materials- detailed in<br>RUSH1FClinical Site<br>Manual of Procedures | Certifiedinvestigatorcoordinator |
| Ocular Exam (includingslit lampbiomicroscopy, indirect ophthalmoscopy and intraocular pressure) | Any equipment is acceptable | Certified investigator |
| Visual Acuity - Refraction | N/A | Clinical site personnel certified for refraction |
| Visual Acuity - ETDRS | EVA system (preferred) otherwise ETDRS charts | Clinical sitepersonnel certified for ETDRS |

| Visual Acuity - LLVA | EVA system (preferred) otherwise ETDRS charts 2.0 neutral density filter to be provided by study | Clinical ste personnebertified for performing ETDRS is also certified to perform LLVA |
|---|---|---|
| Visual Acuity - BRVT | BRVT charts provided by study | Clinical sitepersonnel certified for BRVT |
| Contrast Sensitivity | VectorVision CSV1000E provided by study | Clinical site personned erforming this testing do not require a stud specific certification but must be trained and delegated by the PI per the SSDL |
| SD-OCT | Heidelberg Spectralis | Clinical site personnel certified for SD-OCT |
| Fundus Autofluorescence (on Optos) | Optos (where available) | Clinical sitepersonnel certified for Fundus Autofluorescence on Optos |
| Axial Length and Corneal Curvatur | Any equipment is acceptable | Clinical site personnel performin<br>this testing do notequire a study<br>specific certification but must be<br>trained and delegated by the PI<br>per the SSDL |
| Near Infrared Reflectance Photos | Heidelberg Spectrali(swith 55degree lens) | Clinical site personnel certified for Near Infrared Photos |
| FST | Diagnosys Espion | Clinical site personnel performin<br>this testing do not require a stud<br>specific certification but must be<br>trained and delegated by the PI<br>per the SSDL |
| Static Perimetry | Octopus 900 Pro (GATE Protocol) | Clinical site personnel certified for SP |
| Fundusguided Microperimetry | MAIA | Clinical site personnel certified for MP |
| Kinetic Perimetry (historical) | Any equipment is acceptable | (Historical) Does not need to be<br>performed by study certified<br>personnel or recorded in the<br>RUSH1FStudy Staff Delegation<br>Log |

 $^*$ Required for all sites except with the exception of any site with equivalent equipment approved by the reading observed operations committee.

# Chapter 4: Unanticipated Problems and Adverse Event Reporting

530 4.1 Unanticipated Problems

529

534

535

536

537538

539

540

557

558

559

560

- 531 Site investigators will promptly report to the CC all unanticipated problems meeting the criteria
- below via the Unanticipated Problems eCRTor this protocol, an unanticipated problem is an
- incident, experience, or outcome that mædtthe following criteria:
  - Unexpected(in terms of nature, severity, or frequency) given (a) the research procedures
    that are described in the protocol reladed uments, such as the IRB/Eapproved
    research protocol and informed consent document; and (b) the characteristics of the
    subject population being studied
    - Related or possibly related to participation in the rese(processibly related means there is a reasonable possibility that the incident, experience, or outcome may have been caused by the procedures involved in the research)
- Suggests that the research places participants or others at a greater risk of harm than was previously known or recognize including physical, psychological, economic, or social harm)
- Sites will follow the overseeing IRB's Unanticipated Problem reporting requirements as

  applicable. The CC also will report to the IRB all unanticipated problems not directly involving a
- specific site such as unanticipated problems that occur at the CC or at another participating entity such as a laboratory
- 547 Such as a laboratory
- 548 4.2 Adverse Events
- 549 4.2.1 Definition
- 550 Adverse Event (AE): Any untoward or unfavorable medical occurrence in a human subject,
- including any abnormal sign (for example, abnormal physical exam or laboratory finding),
- symptom, or disease, temporally associated with the subject's participation in the research,
- whetheror not considered related to the subject's participation in the research (modified from the
- 554 definition of AEs in theIntegrated Addendum to ICH E6 (R24)
- Serious Adverse Event (SAE)Any untoward medical occurrence that:
- Results in death
  - Is life-threatening; (a notife-threatening event which, hadbiten more severe, might have become lifthreatening, is not recessarily considered & (S)
  - Requires inpatient hospitalization or prolongation of existing hospitalization
  - Results in persistent or significant disability/incapacity or substantial disruptibe o ability to conduct normal life functions (sight threatening)
- Is a congenital anomaly or birth defect
- Is considered a significant medical event by the investigator based on medical judgment (e.g., may jeopardize the participant or may require medical intervention to prevent one of the outcomes listed above)

#### 566 4.2.2Reportable Adverse Events 567 For this protocol, a reportable includes all events meeting the definition of the above 568 All AEs—whether volunteered by the participant, discovered by stersopnel during 569 questioning, or detected through examination, laboratory test, or other-medialnise reported 570 on an AE form online. 571 The purpose of AE collection for the USH1Fstudy will be to provide historical controls for 572 future clinical trials. As a no greater than minimal risk study, AEs not require any specific 573 reporting to regulatory or oversight bodies. Each Principal Investigator is responsible for abiding 574 by any other reporting requirements specific to his/her IRB or equivalent ethiciabters 575 committee. 576 4.2.3 Relationship of Adverse Event to Study Procedure 577 The study investigator will assess the relationship of Affiny to be related or unrelated to a study 578 procedure by determining if there is a reasonable possibility that Elmeay have been caed 579 by the procedure. 580 To ensure consistency AE causality assessments, investigatoils apply the following general guideline when determining whethe As related: 581 582 Yes 583 There is a plausible temporal relationship between the onset A Etheda study procedure, 584 and the E cannot be readily explained by the participant's clinical state, intercurrent illness, or concomitant therapies; and/or tAE follows a known patterof response to studyprocedure; 585 and/or the AE abates or resolves upon discontinuation study procedure and, if applicable, 586 587 reappears upon rehallenge. 588 No: 589 Evidence exists that the has an etiology other than the procedure (e.g., preexisting medical condition, underlying disease, intercurrent illness, or concomitant medication); and/or 590 591 the AE has no plausible temporal relationship atstudy procedure. 592 4.2.4 Severity (Intensity) of Adverse Event 593 The severity (intensity) of aAE will be rated on a the point scale: (1) mild, (2) moderate, or (3) severeA severity assessment is a clinical determination of the intensity of an eventaThus 594 595 severe E is not necessarily serious. For example, itching for several days may be rated as

- 1. MILD: Usually transient, requires no special treatment, and does not interfere with the participant's daily activities
- 2. MODERATE: Usually causes a low level of inconvenience, discomfort or concern to the participant and may interfere with daily activities but is usually ameliorated by simple therapeutic measures and participant is able to continue in study
- 3. SEVERE: Interrupts a partipant's usual daily activities, causes severe discomfort, may cause discontinuation of study drug, and generally requires systemic drug therapy or other treatment

severe, but may note clinically serious.

596

597

598

599

600

601 602

| 605 | 4.3 Pregnancy Reporting |
|---|---|
| 606<br>607<br>608<br>609<br>610 | If a pregnancy occurs, the participant wellmain in the studyThe occurrence of pregnancy will be reported to the Coordinating Center within se(V) idaysof the site's discovery of the pregnancy (including at screening) the Pregnancy Notification form will be completed within seven(7) calendar daysSites will collect concomitant medications throughout the pregnancy. If an Adverse Event occurs as a result of the pregnancy, then the site will record the Adverse Event on the Adverse Event form. |
| 612 | |
| 613 | |

| 614 | Chapter 5: Miscellaneous Considerations |
|---|---|
| 615 | 5.1 Treatments During the Study |
| 616 | 5.1.1Treatment for PCDH15-Related Retinal Degeneration |
| 617<br>618<br>619<br>620 | Participants <b>enrolled into the final study cohort</b> will be asked to not enroll into experimental treatment trials of underlying conditions related to PCDH15 mutations during the 4-year study duration. Should a participant enroll into a treatment trial during participation, the Executive Committee will decide as to their continuance in RUSH1F. |
| 621 | 5.1.2Treatment for Cystoid Macular Edema |
| 622<br>623 | Participants <b>enrolled into the final study cohort,</b> who need to receive treatment for CME during the study, may continue treatment. |
| 624 | 5.1.3Intraocular Surgical Procedures |
| 625<br>626<br>627<br>628 | Participantsenrolled into the final study cohort who have intraocular surgeduring the study will have follow-up visits timed either before the surgery datates 3 months after the surgery date. Clinical sites ill make reasonable efforts to schedule the participant's follow-up visit as close to the visitargetwindow as possible. |
| 629<br>630 | 5.2 Risks and Benefits |
| 631 | 5.2.1 Risks and Discomforts |
| 632<br>633<br>634<br>635<br>636<br>637<br>638<br>639<br>640 | study will be capturing some information about participants that include identifiable, personal information, like date of birthwill be collected ifpermitted by site's regulatory bodies). The study has procedures in place to protect that information. However, there is a chance that a los of that protection could occur. This would be a loss of confidentiality are are special efforts being made to usure that this does not happen. Otherwise, there are no known risks or discomforts beyond those involved in standard clinical care for patients with retinal degeneration involved in participation in this study, which involves systematically collecting involved in a |
| 641<br>642 | The sections below summarize the risks and discomforts that may be involved in the usual care of the patient during the eriodof prospective data collection. |
| 643<br>644<br>645<br>646<br>647<br>648<br>649<br>650<br>651 | <ul> <li>Risks associated with testing A, KP, SP, Optos FAF, nearinfrared reflectance photos, and PROmay include boredom and frustration, but no lasting adverse effects are associated with these noninvasive tests</li> <li>Dilating eye drops will be used as part of the thalmic examination and before the OCT, FST, and MP. Dilating eye drops may sting, cause lighensitivity, or an allergic reaction. There is a small risk of inducing a narrowgle glaucoma attack from the pupil dilation. However, all participants will have had prior pupil dilation usually on multiple occasions and therefore the risk is extremely small. If glaucoma occurs, treatment is available</li> </ul> |

- IOP ExaminationIn rare instances, the cornea may be scratched during measurement of intra-ocular pressure or use of a contact lens electrode. An abrasidmislikeay be painful, but it heals quickly with no lasting effects a participant experiences a corneal abrasiona tear ointmentary beadministered and an eye patch or gauze may be placed over the eye
  - The risks of genetic testing include emotional psychological stress when patients may learn they have a genetic disease that could be passed along to their children, if information relating to the family, such as adoption and paternity, could be determined from these tests all the genetic testing formation will be kept in confidential laboratory documents and medical records. If data gathered through genetic testing is accidentally released or stolen, it is possible that the information could become available to an insurer, an employer, a relativer someone else. There are discrimination protections in US Federal Law and many State laws, however there is still a small chance that participants could be harmed if a release occurred

#### 666 5.2.2Benefits

- Study participants are not expected to benefit directly fparticipation in this study. Subjects participating in this study may benefit from close attention from the study personnel and PI.
- The risks of participating in the study are outweighed by the benefits including increased
- attention from the study personnel and the ability to contribute to increased understanding
- 671 natural history oPCDH15related retinal degeneration and contribute to future development of
- 672 treatments

657

658 659

660

661

662 663

664

- 5.3 Collection of Pre-Existing Conditions and Medications
- 674 Pre-Existing Condition: Any medical condition that is either present at screening, a chronic
- disease, or a prior condition that could impact the participant's health during the study (e.g., prior
- 676 myocardial infarction or strokevill be recorded.
- Medications: All medication for the treatment of chronic presisting conditions, medical
- 678 conditions, and/oAEs that the participant is currently taking at screening damining the study
- 679 will be recorded Nutraceuticals and preventative that ment also will be recorded.
- 680 5.4 Participant Compensation
- Participant compensation will be specified in t6€.
- 682 5.5 Participant Withdrawal
- Participation in the study is voluntary, and a participant may withdraw at any time. For
- participants who withdraw, their data will be used up utheitime of withdrawal.
- 685 5.6 Confidentiality
- For security and confidentiality purposes, participants will be assigned an identifier that will be
- 687 used instead of their name. Protected health information gathered for this study will be shared
- with the FFB Consortium CC, the Jaeb Center for Health Research in Tampade, USA. De-
- identified participant information may also be provided to research sites involved in the study.

# Chapter 6: Statistical Considerations

The approach to sample size and statistical analyses are summarized below. A detailed statistical analysis plan will be written and finalized prior to the completion of the study. The analysis plan synopsis in this chapter contains the framework of the anticipated final analysis plan.

### 6.1 Sample Size

The sample size evaluation focuses on objective 1 of the study, to characterize the natural history of retinal degeneration associated with biallelic pathogenic mutations in the PCDH15 gene over 4 years on both the structural and functional outcomes of interest. Calculations to address objective 3, explore possible risk factors associated with progression, are summarized. A justification of the selected sample size using percent change for the outcomes of interest is outlined. The precision of the between-eye correlation is also provided.

# 6.1.1 Sample Size Considerations for Evaluating Percent Change from Baseline to 4 Years (All Outcomes)

Longitudinal changes on all outcome parameters being collected will be of interest. Change from baseline to 4 years will be evaluated for sample size purposes. The power/sample size calculations may be used to consider percent change on any outcome measure from baseline to 4 years.

Both eyes of a participant will be assessed for the main outcomes of interest. Thus, if there are N participants, 2N eyes will be available for analysis. However, outcome measures from 2 eyes of a person are typically strongly correlated ( $r \ge 0.5$ ). The contribution of information in this case is (2/(1+r)) instead of 2. Values for the multiplier to the number of participants to obtain an effective sample size are given below:

| r | Effective<br>N |
|-----|----------------|
| 0.0 | 2.00 |
| 0.1 | 1.82 |
| 0.2 | 1.67 |
| 0.3 | 1.54 |
| 0.4 | 1.43 |
| 0.5 | 1.33 |
| 0.6 | 1.25 |
| 0.7 | 1.18 |
| 8.0 | 1.11 |
| 0.9 | 1.05 |
| 1.0 | 1.00 |
- 713 One objective is to estimate the correlation between eyes for the outcome measures; therefore,
- 714 the value of the correlation is not known at the time of study design. We assume here a
- 715 correlation of 0.8. This assumption is conservative in that it requires a higher number of
- 716 participants that other plausible values of r.
- 717 The primary way sample size is evaluated is by considering the precision around the point
- 718 estimates for the outcome measures of interest. Table 1 (including the table of specific values
- 719 corresponding to the graph) provides the half width of the 95% confidence interval (CI) for the
- 720 estimated mean percent change for combinations of the standard deviation (SD) of the
- 721 distribution of percent change and sample size. The larger the SD, the wider the CI, meaning the
- 722 range of possible true values grows.

723

Table 1. Sample size versus half width of 95% confidence interval for the mean percent change for varying standard deviation values

| | Effective Sample Size (N of participants) | | | | |
|---|---|---|---|---|---|
| | n=11 (10) | n= 22 (20) | n= 33 (30) | n= 44 (40) | n=55 (50) |
| SD=20% | 12% | 8% | 7% | 6% | 5% |
| SD=30% | 18% | 13% | 10% | 9% | 8% |
| SD=40% | 24% | 17% | 14% | 12% | 11% |
| SD=50% | 30% | 21% | 17% | 15% | 13% |

- Note: Shaded columns correspond to the range of sample sizes feasible based on preliminary
- 726 patient counts and financial constraints
- 6.1.2Sample Size Considerations for Comparing Percent Change from Baseline to 4 Years
   within Subgroups of Interest (All Outcomes)
- Another important objective for this natural history study will be to explore the association of
- 730 possible risk factors with progression of various functional outcome variables (objective 3).
- 731 Figure 1 considers various expected SDs of the distribution of percent change from baseline to 4
- years per eye and evaluates the power to detect varying differences in average percent change
- 733 from baseline to 4 years, comparing subgroups of various equally distributed sizes. If subgroups
- are not equally sized the detectable difference (with the same power) will be larger. Testing will
- 735 be performed with a Type I ( $\alpha$ ) error rate of 0.05.
- Note: within subgroup point estimates a 6ths will also be important. Table 1 above can be
- applied to potential subgroup sample sizes as well to consider the precision ultabe
- 738 observed.
- 739 Figure 1. Power to conclude there is a difference given varying true difference values,
- 740 population standard deviation, and sample size



Power to conclude there isdifference, when true difference in mean percent changexissx value. Assuming various sample size (subgroups close to equal distribution).

For example, with an effective sample size 22 and an effective sample size of 11 in each group, to have power o80% or more, the true difference needs to be approximately 1.25 SDs (a mean difference of 25% if the SD of the percent change over 4 years 20%). If the effective sample size is 33, the true difference needs to be approximately 1.0 SD (a mean difference SD of the percent change over 4 years is 20%). If the effective sample size is 44, the true difference needs to be approximately 0.86 SDs (a mean difference 17% if the SD of the percent change over 4 years is 20%). Such mean differences are densid large.

# 6.1.3Sample Size Considerations for Precision of the Estimate of the Correlation between Eyes

The intraclass correlation coefficient is used to assess the strength of correlation between eyes. When both eyes have the same mean for the outcome measure, the intraclass correlation coefficient is equal to the standard Pearson correlation coefficient (r). The distribution of r is not symmetric; therefore, CIs for the estimated correlation coefficient are not symmetric. A transformation of r (z = 0.5 \* ln ((1+r)/1-r)) is used to create a variable that is asymptotically

distributed N (0, 1/(sqrt(N-3))) under the null hypothesis that r=0. The table below provides the 95% CI for different estimates of r from the observed data.

#### Table 2. 95% Confidence Intervals for an Observed Value of r

| | N of patients | | | | |
|---|---|---|---|---|---|
| r | n= 10 | n= 20 | n= 30 | n= 40 | n=50 |
| 0.3 | (-0.41,0.78) | (-0.16,0.66) | (-0.07,0.60) | (-0.01,0.56) | (0.02,0.53) |
| 0.4 | (-0.31,0.82) | (-0.05,0.72) | (0.05,0.66) | (0.10,0.63) | (0.14,0.61) |
| 0.5 | (-0.19,0.86) | (0.07,0.77) | (0.17,0.73) | (0.22,0.70) | (0.26,0.68) |
| 0.6 | (-0.05,0.89) | (0.21,0.82) | (0.31,0.79) | (0.35,0.77) | (0.39,0.75) |
| 0.7 | (0.13,0.92) | (0.37,0.87) | (0.45,0.85) | (0.50,0.83) | (0.52,0.82) |
| 8.0 | (0.34,0.95) | (0.55,0.92) | (0.62,0.90) | (0.65,0.89) | (0.67,0.88) |
| 0.9 | (0.62,0.98) | (0.76,0.96) | (0.80,0.95) | (0.82,0.95) | (0.83,0.94) |

Note: Shaded columns correspond to the range of sample sizes feasible based on preliminary patient counts and financial constraints

## 6.1.4Final Sample Size Justification

Longitudinal changes in all outcome parameters being collected will be of interest for objectives 1 and 3. Information on rates of decline for PCDH15, and for inherited retinal degenerations in general, is very limited.

## 770 Data to consider for evaluating sample size:

- Valproic Acid Protocol (VPA) Data (a phase II multiple site, randomized, placebo controlled trial of oral valproic acid for ADRP) [Placebo group N=44; statean be accessed thtps://public.jab.org/ffb/stdy]
  - o Percent Change from Bediene to 1 year, Mean (3):
    - -0.3% (16%) OD
    - -4.9% (17%) OS
- Natural history of 15participants with EYS mutations (McGuigan/Jacobson, 2017)
  - -5.7% per year for VA [8 aprticipants]
  - -5.8% for hnerSegmentOuterSegment (IS/OS\u00abxtent)
- Natural history of 12 participantwith EYSmutations(Miyata/Yoshimura, 2016)
  - -5.2 ±3.1% for IS/OS extent

## 782 Assumptions made:

761

762

765

766

771

772 773

774

775

776 777

778

779780

781

783

784

- Expect average annual decline time PCDH15eyeswill be 5% per year or 02% by 4 years
- True SD of percent change at 4 yeisrlike VPA 1-year SD ofapproximately20%

- 786 If 30 patients or 33 effective eyes are recruited: With an effective sample size of 33, the half
- 787 width of a 95% CI around the point estimate for mean percent change would be 7%. A
- 788 comparison of two equal-sized subgroups would have about 80% power to conclude there is a
- 789 difference if the true difference is 20%.
- 790 If 40 patients or 44 effective eyes are recruited: With an effective sample size of 44, the half
- 791 width of a 95% CI around the point estimate for mean percent change would be 6%. A
- 792 comparison of two equal-sized subgroups would have about 80% power to conclude there is a
- 793 difference if the true difference is 17%.
- For objective 4 of evaluating variability and symmetry, a sample size of 30 participants for
- 795 Vision Cohorts 1 and 2 will have a 95% CI of (0.17,0.73) when observed r equals to 0.5, and
- 796 (0.62,0.90) when observed r equals to 0.8. A sample size of 40 participants for Vision Cohorts 1
- 797 and 2 will have a 95% CI of (0.22,0.70) when observed r equals to 0.5, and (0.65,0.89) when
- 798 observed r equals to 0.8.
- Recruitment is anticipated to take 10 months from the time of study launch.
- 800 6.2 Data Analysis

807

808

809 810

811

812

813

814

815

816

817

818

819

820

821

822

823

824

825

826

- The analysis plans below are written with respect to the majority of outcomes of interest.
- 802 Analyses will include data on both eyes for each participant, and confidence intervals will adjust
- 803 for correlation between 2 eyes of the same participant.
- 804 6.2.1 Primary Objectives Analyses
- The primary objectives of the natural history study and brief analysis plan for each are as follows.
  - Characterize the naturalishory of retinal degeneration associated with biallelic disease causing variants in the PCDH15 gene over 4 years, as measured using functional, structural, and patienteported outcommeasures
    - a. Analysis planfor functional and structural measur she distribution of each outcome at each visit will be summarized (including tabulating categorically, as well as means Ds medians, quartiles, ranges; both the absolute change and percent change will be evaluated sts performed multiple times will banalyzed using average of all available tests determine the average annual rate of progression in the population for each outcome, a repeated measure least squares regression model will be fit using all available outcome data at baseline and all annual visits. Multiple imputation will be used to impute the outcome values for all missing time points (including participants who discontinue follow up prior to 48 months). Secondary analyses using binary definitions of outcome measures will also be explored in time to event analyses; Kap lateier estimates with 95% confidence intervals will be calculated
    - b. Analysis plan for PRO measures he scoring of each questionnaire will be completed according to the procedures for each instrument and is detailed further in a separate statistical analysis plan. Baseline scores will be cross tabulated with categorical (severity of disease) versions of the outcome measures of interest at baseline. Changes in scores will be cross tabulated with binary (progression of disease) versions of the outcome measures of interest at the 24- and 48-month

| 828<br>829 | visits. A generalized linear model adjusted for baseline differences will be explored. | |
|---|---|---|
| 830<br>831<br>832 | <ol> <li>Explorewhether structural outcome measures can be validated as surrogates for<br/>functional outomes in individuals with biallelic pathogenic mutations in PMDH15<br/>gene</li> </ol> | |
| 833<br>834<br>835 | <ul> <li>a. <u>Analysis plan</u> Scatterplots and Spearman correlation coefficients of chang<br/>SD-OCT EZ area versuls progression from baseline to each visit will be<br/>evaluated.</li> </ul> | es in |
| 836<br>837<br>838 | 3. Explorepossible risk factors (genotype, phenotype, environmental, and comorbidit for progression of the outcome measures at 4 years in individuals with biallelic pathogenic mutations in the CDH15gene | ies) |
| 839<br>840<br>841<br>842<br>843 | <ul> <li>Analysis plan The distribution of each outcome in terms both absolution change and percent change from baseline to 4 years will be sum (including tabulating categorically, as Iwas means, standard deviation medians, quartiles), stratified by categorical levels of each potential rise of interest(listed below). Potential riskfactors to evaluate include:</li> </ul> | marized<br>ons, |
| 844 | o Phenotypic: | |
| 845<br>846<br>847<br>848<br>849<br>850<br>851<br>852<br>853<br>854<br>855<br>856<br>857<br>858 | <ul> <li>Clinical diagnosis</li> <li>Age of onset ofnitial vision symptoms</li> <li>Gender</li> <li>Race/ethnicity</li> <li>Visual acuity</li> <li>Lens Status (phakic/pseudophakic/aphakic)</li> <li>SD-OCT (as factors related to SP Hill Øfsion (HOV)) <ul> <li>Presence of cysts</li> <li>Central subfield thickness</li> </ul> </li> <li>MP <ul> <li>Mean retinal sensitivity</li> </ul> </li> <li>SP (as factors related &amp;D-OCT EZ area) <ul> <li>Volume of 30 degrees HOV</li> <li>Mean sensitivity</li> </ul> </li> </ul> | |
| 861<br>862 | <ul><li>Full field HOV</li><li>Genotypic:</li></ul> | |
| 863 | • Characterizations of the variants on the <i>PCDH15</i> protein | |
| 864 | <ul> <li>Environmental factors</li> </ul> | |
| 865<br>866<br>867<br>868 | <ul> <li>Smoking status at baseline</li> <li>Vitamin A use at baseline</li> <li>Docosahexaenoic acid (DHA) use at baseline</li> <li>Lutein use at baseline</li> </ul> | |

- 4. Evaluate variability of repeat perimetry testing of symmetry of left and right eye outcomes over 4 years in individuals with biallelic pathogenic mutations PACD#15 gene
  - a. <u>Analysis plan for variability of repeat perimetry testing at baseline:</u> Scatterplots and Spearman correlation coefficients for pairs (first versus second) of testing values for each repeated perimetry test. Bland-Altman plots of difference versus the mean value will be inspected. The intraclass correlation coefficient of the values and the within-person variance will be estimated.
  - b. Analysis plan for the symmetry of left eye versus right eye: At baseline and each subsequent testing time, the symmetry of the test result values from the left and right eyes will be assessed and the symmetry of the change from baseline from the left and right eyes will be assessed for each follow-up visit. Bland-Altman plots of the inter-eye difference versus the mean value will be inspected. The intraclass correlation coefficient of the values will be estimated.

## 6.2.2Interim Data Analysis

No formal interim analysis or "stopping guidelines" are planned for determining early stopping according to statistical rules, as no intervention is being studied and thus early efficacy and safety signals are not applicable.

Interim analyses will be planned for other reasons, including to evaluate data at baseline and annual visits for reporting in preliminary manuscripts, as well as monitoring data for recruitment and retention benchmarks, and quality assurance throughout the duration of the study. The FFB Consortium Executive Committee will review and oversee these data and their use in reporting.

| 892 | Chapter 7: Data Collection and Monitoring |
|---|---|
| 893 | 7.1 Case Report Forms and Other Data Collection |
| 894<br>895<br>896<br>897<br>898<br>899<br>900 | The main study data are collected electronic case report formsQRFs) When data are directly collected in GRFs this will be considered the source dafter any data points for which the eCRF is not considered source (death results which are transcribed from a printed report into the eCRF), the original source documentations be maintained the participant's study chart or medical record his source must be readily verifiable against the values entered into eCRF. Even where all study data are directly entered into the eCRdffscet visits, evidence of interaction with a live subject must be recorded (e.g., office note, visit record, etc.) and provided to the coordinating center for review |
| 902<br>903<br>904 | The Central Lab will generate genetic reports from retinal dystroph genetic pael testing and or family member testing nalysis as applicable. These reports will be uploaded to the FFB Consortium study website and made available to the clinical site. |
| 905<br>906<br>907<br>908<br>909 | The CGA will review the genetic lab rep(xx) submitted by the clinical site during enetic screening against the genetic eCRF data to ensure that the data entered by the clinical site are consistent with the sour(xx) provided prior to the Baseline visit he CGA will document his/her verification of these genetic data on the FFB Coting or study website and the clinical site will be notified of the results of the review. |
| 910<br>911<br>912<br>913 | In addition to providing interpretation/evaluation of whether or not PPGDH15 mutations are causative of the disease the FFB Consortium study webs tree section 2.4.2), the Genetics Committee will review and provide approval for the use of genetic reports from search labs to be use for determining participant eligibility. |
| 914<br>915<br>916<br>917 | Reading Centerwill conduct grading ofhe study data collected for M8D-OCT, Optos FAF, and SPusing the FFB Consortium study website Reading Center will conduct quality review only of the first ERG obtained from each inical site using the FFB Consortium study website. These data will remain in the study database and will not be provided to the clinical site. |
| 918<br>919<br>920<br>921 | Each participating site will maintain appropriate medical and research records for this trial, in compliance with International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (CH) E6 and regulatory and institutional requirements for the protection of confidentiality of participants. |
| 922 | 7.2 Study Records Retention |
| 923<br>924<br>925<br>926<br>927 | Study documents/ill be retained for a minimum of x (6) years from the daten which the CC receives IRB approval to close the studly ese documents/ill be retained for a longer period, however, if required by local regulations. No records will be destroyed without the written consent of the C. It is the responsibility of the C to inform the investigator wheat udy documents no longer need to be retained. |
| 928 | 7.3 Quality Assurance and Monitoring |
| 929<br>930<br>931 | Designated personnel from the will be responsible for maintaining quality assurance (QA) and quality cotrol (QC) systems to ensure that the clinical portion of the trial is conducted and data are generated, documented and reported in compliance with the protocol, GCP and the |

- 932 applicable regulatory requirements well as to ensure that the rights and wiellipef trial 933 participants are protected and that the reported trial data are accurate, complete, and verifiable Consistent with Integrated Addendum t6H E6 (R2<sup>94</sup>, arisk-based monitoring (RBM) plan 934 will be developed and revised as neededngthe study This plan describes in detail who will 935 936 conduct the monitoring, at what frequency monitoring will be done, at what levelable det 937 monitoring will be performed, and the distribution of monitoring reports. 938 As much as possible, remote monitoring we performed in reatime with onsite monitoring 939 performed to evaluate the verity and completeness of the key site data. Elements of the RBM planmay include: 940 941 Qualification assessment, training, and certification for sites and site personnel 942 Oversight IRB/EC coverage and informed consent procedures 943 • Central (remote) data monitoring: validation of data entry, data edits/audit trail, protocol review of entered data and edits, statistical monitoring, study closeout 944 • On-site monitoring (site visits): sourcdata verification, site visit report 945 946 Communications with site staff 947 Participant retention and visit completion 948 Quality control reports 949 Management of noncompliance 950 Documenting monitoring activities 951 AE reporting 952 CC representatives or their designees mist the study facilities at any time in order to maintain current and personal knowledge of the study through review of the records, comparison 953 954 with source documents, observation and discussion of the conduct and progress of the study. 955 investigationabite will provide direct access to all trial related sites, source data/documents, and reports for the purpose of monitoring and auditing by the sponsor, and inspection by local and 956 957 regulatory authorities. 958 7.4 Protocol Deviations 959 A protocol deviation is anyoncompliance with the clinical trial protocol, GCP, or procedure 960 requirements. The noncompliance may be either on the part of the participant, the investigator,
- or the study site staff. As a result of deviations, corrective actions are to be developed itey

962

- 963 The site Plandstudy staffdelegated to study responsibilities responsible for knowing and
- adhering to their IREC requirements.

and implemented promptly.

| 965 | Chapter 8: Ethics/Protection of Human Participants |
|---|---|
| 966 | 8.1 Ethical Standard |
| 967<br>968<br>969 | Theinvestigator will ensure that this study is conducted in full conformity with Regulations for the Protection of Human Participants of Research codified in the Conformity with Regulations (CFR) Part 46, 21 CFR Part 50, 21 CFR Part 56, and/or the ICH E6. |
| 970 | 8.2 Institutional Review Boards and Ethics Committees |
| 971<br>972<br>973<br>974<br>975<br>976 | The protocolJCF(s), recruitment materials, and all participant materials will be submitted to the IRB or EC for review and approval. Approval of both the protocol and the obtained before any participant is enrolled. Any amendment to the protocol will require review and approval by the IRB EC before the changes are implemented to the studychalles to the consent form will be IRB ECapproved; a determination will be made regarding whether previously consented participants need to be presented. |
| 977 | 8.3 Informed Consent Process |
| 978 | 8.3.1 Consent Procedures and Documentation |
| 979<br>980<br>981<br>982<br>983<br>984<br>985<br>986<br>987<br>988<br>989 | Informed consent is a processat is initiated prior to the individual's agreeing to participate in the study and continues throughout the individual's study participation. All consent forms will be IRB-or EC approved and the case of written consettine participant will begiven the opportunity to carefully eadand review the document. For any form of consentresented (written or verbal), the investigatoor his/her designe (as approved by the IRB/EQ) ill explain the research study to the participant and answer any questions ay arise. All participants will receive a verbal explanation in terms suited to their comprehension of the purposes, procedures, and potential risks of the study and of their rights as research participatents ive discussion of risks and posteribenefits of participation will be provided to the participants and their families. Participants will be asked o carefully consider the consent form presented to themandhave anyquestions answered prior to signing. |
| 990<br>991<br>992<br>993<br>994<br>995 | Participantswill have the opportunity to discuss the study with their surrogates or think about it prior to agreeing to participant articipants must sign the CF prior to any procedures being done specifically for the stud articipants may withdraw consent at any tenthroughout the course of the trial. A copy of the F will be given toparticipants for their records. The rights and welfare of participants will be protected by emphasizing to them that the quality of their medical care will not be adversely affectethey decline to participate in this study. |
| 996 | 8.3.2Participant and Data Confidentiality |
| 997<br>998<br>999<br>1000<br>1001<br>1002 | Participant confidentiality is strictly held in trust by the participating investigators, their staff, the funder(s) and their agents. This confidentiality is extender genetic tests in addition to the clinical information relating to participants. Therefore, the study protocol, documentation, data, and all other information generated will be held in strict confidence. No information concerning the tudy, or the data will be released to any unauthorized third party without prior written approval of the sponsor. |

| 1003<br>1004<br>1005<br>1006<br>1007 | The CC, other authorized endors or epresentatives of the IRBs/ECs or regulatory agencies ay inspect all documents and or eds required to be maintained by the investigator, including but not limited to medical records (office, clinic, or hospital) for the participants in this study. The clinical study site will permit access to such records. |
|---|---|
| 1008<br>1009<br>1010<br>1011 | The study participant's contact information will be securely stored at each clinical site for internal use during the study. At the end of the study, all records will continue to be kept in a secure location for as long a period as dictatetheyeviewingRB/EC, institutional policies, or sponsor requirements |
| 1012<br>1013<br>1014<br>1015<br>1016<br>1017<br>1018<br>1019 | Study participant research data, which is for purposes of statistical analysis and scientific reporting, will be transmitted to and stored at HTHE ConsortiumCC, located at the Jaeb Center for Health Research in Tampa, FloridThis will not include the participant's contact or identifying information unless otherwise specified in the informed consent.formathera unique study identification number will identify individual participants and their research data The studydata entry and study management systems used by clinical sites the TEP ConsortiumCC research staff will be secured and password protected. At the end of the study, all study databases will be detentified and archived at the TEP ConsortiumCC. |
| 1020 | 8.4 Stored Specimens |
| 1021<br>1022<br>1023<br>1024<br>1025 | With the participant's approval and as approved by the IRB/ECs, deidentified biological samplescollected for genetic testing screening groups B and will be stored a Blueprint Genetic suntil the FFB Study Team notifies them in wirg to destroy the samples. We expect the samples to be destroyed (1) year after the end of the study. |

### 1026

# Chapter 9: References

- Zrada SE, Braat K, Doty RL, Laties AM. Olfactory loss in Usher syndrome: Another sensory deficit? AmJ Med Genet1996;64(4):602603.
- Petit C. Usher Syndrome: From Genetics to Pathoger Rev Genomics Hum Genet.2001;2(1):271297.
- Fakin A, JareVidmar M, Glavac D, Bonnet C, Petit C, Hawlina M. Fundus autofluorescence and optical coherencedomaphy in relation to visual function in Usher syndrome type 1 and 2sion Res2012;75:6070.
- 1034 4. Pakarinen L, Tuppurainen K, Laippala P, Mäntyjärvi M, Puhakka H. The ophthalmological course of Usher syndrome typelnlil. Ophthalmol. 1995;19(5):307 311.
- 1037 5. Ness SL, BerYosef T, BarLev A, et al. Genetic homogeneity and phenotypic variability among Ashkenazi Jews with Usher syndrome type Med Genet2003;40(10):767.
- Ahmed ZM, Riazuddin S, Ahmad J, et al. PCDH15 is expressed in the neurosensory epithelium of the eye and ear and mutant alleles are responsible for both USH1F and DFNB23. Hum Mol Genet2003;12(24):321\foxbar{2}223.
- 5. Schietroma C, Parain K, Estivalet A, et al. Usher syndrome typessociated cadherins shape the photoreceptor outer segmetall Biol.2017;216(6):1849/864.
- 1044 8. Ahmed ZM, Riazuddin S, Aye S, et al. Gene structure and mutant alleles of PCDH15: nonsyndromic deafness DFNB23 and type 1 Usher syndidome.Genet. 2008;124(3):215223.
- Theng QY, Yan D, Ouyang XM, et al. Digenic inheritance of deafness caused by mutations in genes encoding cadherin 23 and protocadherin 15 in mice and humans. Mol Gen.2004;14(1):103111.
- 1050 10. Ben-Yosef T, Ness SL, Madeo AC, et al. A Mutation of PCDH15 among Ashkenazi Jews with the Type 1 Usher Syndrom Lengl J of Med2003;348(17):664-1670.
- 1052 11. Jacobson SG, Cideciyan AV, Aleman TS, et al. Usher syndromes due to MYO7A, PCDH15, USH2A or GPR98 mutations share retinal disease mechahism/Mol Genet 2008:17(15):240 2415.
- 1055 12. Stingl K, Kurtenbach A, Hahn G, et al. F-filleld electroretinography, situal acuity and visual fields in Usher syndrome: a multicentre European s Dodg. Ophthalmol. 2019;139(2):154160.
- 1058 13. Rebibo-Sabbah A, Nudelman I, Ahmed ZM, Baasov T, Browsef T. In vitro and ex vivo suppression by aminoglycosides of PCDH15 nonsensætionus underlying type 1 Usher syndromeHum Genet2007;122(34):373-381.
- Birch DG, Locke KG, Felius J, et al. Rates of decline in regions of the visual field defined by frequencylomain optical coherence tomography in patients with RPGR mediated Xlinked retinitis pigmentos © phthalmology 2015;122(4):83 3839.
- Hariri AH, Zhang HY, Ho A, et al. Quantification of Ellipsoid Zone Changes in Retinitis Pigmentosa Using en Face Spectral Dom@iptical Coherence TomographJAMA
  Ophthalmology2016;134(6:628-635.
- 1067 16. Han RC, Gray JM, Han J, Maclaren RE, Jolly JK. Optimisation of dark adaptation time required for mesopic microperimetry J Ophthalmol2019;103(8):1092.

- 1069 17. Stingl KT, Kuehlewein L, Weisschuh N, et al. Chromatic #Füeld Stimulus Thresdrid and Pupillography as Functional Markers for Latege, EarlyOnset Retinitis Pigmentosa Caused by CRB1 Mutationsansl Vis Sci Techno2019;8(6):4545.
- 1072 18. Birch DG, Cheng P, Duncan JL, et al. The RUSH2A Study:-**Best**ected Visual Acuity, Full-Field Electroretinography Amplitudes, and **Full**eld Stimulus Thresholds at BaselineTransl Vis Sci Techno2020;9(11):99.
- 1075 19. Bennett LD, Klein M, Locke KG, Kiser K, Birch DG. Darkdapted Chromatic 1076 Perimetry for Measuring Rod Visual Fields in Patienitts Retinitis Pigmentosa Transl 1077 Vis Sci Technol 2017;6(4):1515.
- 1078 20. Jacobson SG, Voigt WJ, PareMJ et al. Automated Lightand Dark Adapted Perimetry for Evaluating Retinitis Pigmentos@phthalmology.1986;93(12):16041611.
- 1080 21. Stingl K, Nowomiejska K, Kuehlewein L, et al. Clinical protocols for the evaluation of rod function.Ophthalmologica2020.
- 1082 22. Kelbsch C, Stingl K, Kempf M, et al. Objective Measurement of Local Rod and Cone 1083 Function Using Gaz©ontrolled Chromatic Pupil Campimetry in HealtBubjects. 1084 Transl Vis Sci Techno2019;8(6):1919.
- 1085 23. Rare diseases: Natural History Studies for Drug Development: Guidance for Industry, Draft Guidance. In: U.S Department of Health and Human Services Food and Drug Administration. ed2019.
- 1088 24. Integrated Addendum to ICH E6 (R1): Guideline for Good Clinical Practice: E6(R2). In: U.S. Department of Health and Human Services Food and Drug Administration, ed2016.